CLINICAL TRIAL: NCT02599025
Title: Effect of Posture and Passive Cycling on Cardiac Autonomic Control System in Children With Severe Cerebral Palsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ziv Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: ziv-0089015
Record Dates: First submitted 2015-11-04; First posted 2015-11-06 (Estimated); Last update posted 2015-11-06 (Estimated); Status verified 2015-11

CONDITIONS: Cerebral Palsy
Keywords: Cerebral palsy; passive cycling; autonomic control system
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Supine position (No Intervention): Children tested while lying down
- Standing position (No Intervention): Children tested while standing
- Cycling supine postion (Experimental): Children lying down with APT cycling system
  Interventions: Device: APT cycling system
- Cycling standing postion (Experimental): Children standing with Innowalk cycling system
  Interventions: Device: Innowalk cycling system

INTERVENTIONS:
Device: Innowalk cycling system — Innowalk is a unique, motorized medical device
  Arms: Cycling standing postion
Device: APT cycling system — APT is used as a rehabilitative device that cycles the feet automatically or by the individual
  Arms: Cycling supine postion

SUMMARY:
The investigators will examine the immediate contribution of position and movement on the functioning of the autonomic cardiac control system.

DETAILED DESCRIPTION:
Standing position is a routine therapeutic tool for improving bone density in children with cerebral palsy. The autonomous immediate response for these children is defective. In recent years it has been shown that there is an association between bone density and autonomic function .

In this paper the investigators will examine how the addition of movement to standing subjects contribute to changes in heart rate and blood pressure.

The hypothesis is that the integration of movement while standing presents a change in the autonomic response and thus may improve bone density.

ELIGIBILITY:
Inclusion Criteria:

* Motor ability of GMFCS IV-V

Exclusion Criteria:

* Children with hip subluxation
* On Baclofen inhaler treatment
* Heart disease
* surgical procedures

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Estimated)
Dates: Start 2016-02; Primary Completion 2017-02 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Heart rate variability | 10 minutes each position
Blood pressure monitoring | 10 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Luder, MD, Principal Investigator — Ziv Medical Center, Zefat